CLINICAL TRIAL: NCT00736021
Title: Post-marketing, Twelve Weeks, Open Label Study of up to 40 mg. Escitalopram in Chronic PTSD
Brief Title: Treatment of Post-traumatic Stress Disorder With High Doses of Escitalopram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arieh Y. Shalev, M.D., Department of Psychiatry, Hadassah University Hospital, Jerusalem, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO_SHALEV_02
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2008-09

CONDITIONS: Stress Disorders, Post Traumatic
Keywords: PTSD; Pharmacological Treatment; SSRI; Escitalopram; Anxiety Disorders
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Single arm (open label study): Provide twelve weeks of treatment with high does (40 mg daily) of escitalopram to trauma survivors with chronic PTSD.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Up to 40 mg oral dose in 10 or 20 mg tablets taken twice daily
  Other Names: Lexapro, Cipralex

SUMMARY:
The study evaluates the hypothesis that large doses of Escitalopram will reduce symptoms of chronic post-traumatic stress disorder (PTSD) in adult civilian survivors of traumatic events.

Forty survivors of carefully documented traumatic events who had been followed for more than two years and have not improved will receive up to 40 mg of Escitalopram (daily) for twelve weeks

Symptoms of PTSD, depression, anxiety disorders, quality of life and global clinical impression, as well as emergent side effects will be recorded every two weeks (one week for the first four weeks.

The primary outcome measure will be symptoms of PTSD as recorded at the end of the study (or the last meeting with the patient - Last Observation Carried Forward).

The secondary outcome criteria will be treatment continuation, as expressed in the proportion of patients leaving the study for either lack of effect or side effects.

DETAILED DESCRIPTION:
The study evaluates the hypothesis that large doses of Escitalopram will reduce symptoms of chronic post-traumatic stress disorder (PTSD)

Forty adult survivors of carefully documented traumatic events who had been followed for more than two years and have not improved will receive up to 40 mg of Escitalopram (daily) for twelve weeks

Symptoms of PTSD, depression, anxiety disorders, quality of life and global clinical impression, as well as emergent side effects will be recorded every two weeks (one week for the first four weeks.

The primary outcome measure will be symptoms of PTSD as recorded at the end of the study (or the last meeting with the patient - Last Observation Carried Forward).

The secondary outcome criteria will be treatment continuation, as expressed in the proportion of patients leaving the study for either lack of effect or side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult survivors of traumatic events with chronic PTSD

Exclusion Criteria:

* Individuals with past history of psychotic disorder, bipolar disorder, opiate or stimulants abuse.
* Individuals currently on anti-depressant therapy.
* Individuals with past history of a failure to respond to escitalopram
* Pregnant Women
* Medical condition excluding the treatment with escitalopram (e.g., renal or hepatic insufficiency). Current, life threatening medical illness. History or severe side effects with escitalopram (e.g., hyponatremia)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder (PTSD) and PTSD symptoms as recorded by the Clinicians Administered PTSD Scale (CAPS) | Twelve Weeks on Active Medication

SECONDARY OUTCOMES:
Proportion of Participants completing the study | twelve weeks of active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Areh Y SHALEV, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel